CLINICAL TRIAL: NCT03209141
Title: Impedance Cardiography in the Evaluation of Left Ventricular Diastolic Dysfunction in Patients With Arterial Hypertension Study (IMPEDDANS)
Brief Title: Screening of Diastolic Dysfunction With Impedance Cardiography in Hypertensive Patients
Acronym: IMPEDDANS
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Responsible Party: Sponsor
Other Study IDs: CHLC.CI.165.2013
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Hypertension; Diastolic Dysfunction
Keywords: hypertension; Diastolic Dysfunction; impedance cardiography; echocardiography
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diastolic dysfunctional hypertension: Patients with confirmed arterial hypertension and diastolic dysfunction by echocardiographic diastolic function evaluation
  Interventions: Diagnostic Test: Diastolic function evaluation
- Non diastolic dysfunctional hypertension: Patients with confirmed arterial hypertension and without diastolic dysfunction by echocardiographic diastolic function evaluation
  Interventions: Diagnostic Test: Diastolic function evaluation

INTERVENTIONS:
Diagnostic Test: Diastolic function evaluation — Diastolic function assessed by impedance cardiography (test to be validated) is compared with the assessment by echocardiography (clinical standard)

SUMMARY:
Arterial hypertension (AHT) is responsible for important morbidity and mortality. The cardiac repercussion of AHT is usually assessed by electrocardiography and echocardiography, time-consuming, technically demanding examinations that require experienced operators, which limits their use for screening diastolic dysfunction. Alternative tools for the screening of diastolic function in hypertensive patients are needed. Impedance cardiography (IC) is presently used in the study of AHT and in the optimization of antihypertensive therapy. It seems an attractive and economical option to change the clinical approach for screening; however, its validation in well-defined populations is required to sustain its use in clinical practice. The IMPEDDANS study aims to validate IC for screening left ventricular diastolic dysfunction in outclinic patients with AHT, using functional echocardiography as the clinical standard. Descriptive and analytical study with analysis of the agreement between the diagnosis of diastolic dysfunction and its degree, as well as the parameters obtained by impedance cardiography and echocardiography in patients with AHT.

DETAILED DESCRIPTION:
BACKGROUND. Impedance cardiography (IC) is a complementary diagnostic test used in the study of arterial hypertension (AHT) and in the optimization of antihypertensive therapy. It is easy-to-execute, non-operator-dependent and cost-effective. It analyses and registers hemodynamic changes through the measurement of electrical resistance changes in the thorax and translates them graphically as impedance and electrocardiogram waveforms. IC has evolved in recent years, making it an attractive and economical tool, particularly in screening settings and there is extensive published literature on its usefulness. More widespread use of IC has been limited due to limitations of the studies, mostly cross-sectional, with small samples, recruiting hemodynamically stable patients and providing inconsistent estimates of accuracy and reproducibility in different settings.

AHT is responsible for high morbidity and mortality. In Portugal, according to PHYSA study, has overall prevalence of hypertension, in 2014, of 42.2% (44.4% in men, 40.2% in women). The progression of hypertensive heart disease involves myocardial fibrosis and changes in left ventricular geometry that precedes functional changes. Diastolic dysfunction is part of this continuum, and despite the growing recognition of its importance, it is generally undervalued because of the difficulty in its diagnosis and the absence of effective therapies. This reinforces the importance of finding alternative tests that provide important information for an initial assessment of diastolic function in hypertensive patients.

This study intends to define the importance and usefulness of IC in the evaluation of LV diastolic dysfunction in patients with AHT.

METHODS. Study Design. This is a validation study of a diagnostic method used in a new context, comparing it with the diagnostic method currently used for this effect in usual clinical practice. Its purpose is to determine the positive predictive value, negative predictive value, sensitivity and specificity of the presence of the D wave, the isovolumetric relaxation time, the systolic time ratio (STR) and thoracic fluid content (TFC) by IC, for the diagnosis of LV diastolic dysfunction (LVDD). To study the relationship between LV geometry, hemodynamic profile, diastolic dysfunction and its degree (confirmed by echocardiography) in hypertensive patients with diastolic dysfunction. We chose to perform a concordance study between IC and echocardiography, the validated , non-invasive test used for the clinical diagnosis of LVDD as well as for the characterization of hypertensive cardiopathy.

To calculate the sample size we considered the primary endpoint (concordance of the diagnosis of diastolic dysfunction between IC and echocardiography). Thus, considering a hypothesized positive predictive value of 70 ± 5% of the parameters obtained by IC, 77 individuals are estimated to be able to verify the expected positive predictive value with 95% confidence. Since the prevalence of diastolic dysfunction in patients with AHT estimated to be approximately 50% in most studies, the sample size is doubled for 154 hypertensive patients.

Evaluation. Participants will be systematically assessed by IC and echocardiography, with a maximum interval of 8 days between them, to obtain the parameters to be used in the validation and concordance studies. To ensure that both tests are performed under similar conditions, evaluations matching variations greater than 10% in BP or variations in excess of 5% in HR will not be considered. These patients should, if possible, repeat one of the exams. If they maintain variations greater than those defined, they should be excluded from the study.

Baseline Data. Ambulatory clinic protocol for patients followed for AHT require clinical evaluation, blood test, electrocardiogram and, eventually, 24 hours ambulatory blood pressure monitoring (AMBP). Data regarding the comorbidities and pharmacotherapy will be collected. Anthropometric data regarding adiposity and vital signs will be registed and body mass index calculated as weight (kg) divided by height (m) squared. Blood pressure will be measured in a quiet room with semiautomatic device (Omron HEM-907XL, Omron Healthcare, Bannockburn, Illinois, USA) with an appropriate cuff according with the established recommendations. If necessary 24 hours ABPM will be performed using an ABPM device - Spacelabs model 90207 (Issaquah, Washington, USA) also according with current guidelines. Electrocardiogram will be performed per institutional protocol with a Page Writer TC 30, Philips, Eindhoven, Netherlands. The analytical screening evaluation includes complete blood count, haematocrit, urinalysis, urine microalbumin, serum sodium, potassium, creatinine (estimated or measured glomerular filtration rate [GFR]), and calcium, uric acid, glycated haemoglobin, lipid profile following a 9- to 12-hour fast (total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, and triglycerides), thyroid-stimulating hormone and brain natriuretic peptide.

Impedance Cardiography. Impedance cardiography will be carried out in a single centre by a cardiopneumology technician with Niccomo continuous cardiac output monitor (Medis, GmbH, Ilmenau, Germany). This equipment uses the technique of four electrodes, two of current application and two others that detect the changes of voltage. As the current amplitude is constant, the voltage detected is proportional to the tissue impedance. Patients must present with fasting of 6 hours but must take their antihypertensive drugs and the examination is carried out in 4 phases after an initial 5 minutes hemodynamic stabilization period: 1. supine position I - 20 minutes continuous recording; 2. 70º orthostatism -with the help of the tilting table for 10 min in continuous recording; 3. tilt-back at 0º; 4. supine position II - 10 min continuous recording. The examination is interrupted if there is syncope or pre-syncope; dizziness, nausea and malaise associated with poorly tolerated hypotension and / or bradycardia; pain / precordial discomfort; ECG ST segment changes; Systolic blood pressure > 210mmHg.

Transthoracic Echocardiography. Transthoracic echocardiography will be performed in Vivid E9 and S5 devices (GE Healthcare, Chicago, Illinois, USA) by experienced cardiologists. The exam will be held in the echocardiography laboratories of two reference centers. To ensure uniformity of evaluation and correct evaluation all exams will be reviewed by a second cardiologist with experience in the technic. In order to define and grade diastolic dysfunction will be recorded left atrium volume index, the velocities E, A, septal e´, lateral e´, deceleration time (DT), isovolumetric relaxation time (IRVT), atrial reverse velocity (Ar) and E/A ratio variation with Valsalva maneuver (last two will only valued if the patient cooperates and if the images obtained have the necessary quality for analysis) as recommended by 2009 guidelines. Left ventricular geometry will be defined accordingly with international recommendations.

Analytic Statistics. The diagnostic validity parameters will be calculated with 95% confidence intervals, using logistic regression models. The positive and negative predictive values will be calculated and the sensitivity and specificity will be estimated; receiver-operator curves (ROC) will also be analysed, with the calculation of the area under the curve. Diagnostic models with more than one parameter will be tested, using multivariable analysis, logistic and linear regression. For the analysis of agreement between the parameters obtained by ICG and echocardiography, the Bland-Altman method will be used with STATA® and R-project® software.

ELIGIBILITY:
Inclusion Criteria:

* grade 2 or 3 hypertension (systolic blood pressure ≥ 160 mmHg and/or with diastolic blood pressure values ≥ 100 mmHg) and/or with resistant hypertension (as defined by European Society of Cardiology

Exclusion Criteria:

* pregnancy,
* height less than 120 cm or more than 230 cm,
* weight less than 30 kg or greater than 155 kg,
* heart failure II-IV NYHA,
* heart rate (HR) less than 50 bpm or greater than 110 bpm,
* atrial fibrillation or flutter,
* > 3 premature ventricular contractions per hour,
* complete left bundle branch or atrioventricular block,
* severe valvulopathies,
* constrictive pericarditis,
* hypertrophic and restrictive cardiomyopathy,
* prior history of ischemic heart disease and/or segmental kinetics alterations assessed by echocardiography,
* left ejection fraction < 50%,
* poor echocardiographic window ,
* pacemaker.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with arterial hypertension attending the outpatient clinic consultation
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Predictive value of impedance cardiography to identify diastolic dysfunction | Less than 10 days between measurements
  Positive predictive value of impedance cardiography to identify diastolic dysfunction, compared with echocardiography
Area under the curve (AUC) | Less than 10 days between measurements
  The area under the receiver-operator curves (ROC) for identification of diastolic dysfunction by impedance cardiography, compared with echocardiography

SECONDARY OUTCOMES:
Negative predictive value of impedance cardiography to identify diastolic dysfunction | Less than 10 days between measurements
  Negative predictive value of impedance cardiography to identify diastolic dysfunction, compared with echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo N Leão, MD, Principal Investigator — Centro Hospitalar de Lisboa Central
Locations (3):
- Portugal (3):
  - Consulta de Hipertensão Arterial, UF Medicina 1.4 do Hospital São José, Centro Hospitalar de Lisboa Central, Lisbon
  - Consulta de Risco Vascular da Unidade Funcional Medicina 1.2, Hospital São José, Centro Hospitalar de Lisboa Central, Lisbon
  - Núcleo de Hipertensão Arterial, Consulta de Medicina do Hospital de Santa Marta, Centro Hospitalar de Lisboa Central, Lisbon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ventura HO, Taler SJ, Strobeck JE. Hypertension as a hemodynamic disease: the role of impedance cardiography in diagnostic, prognostic, and therapeutic decision making. Am J Hypertens. 2005 Feb;18(2 Pt 2):26S-43S. doi: 10.1016/j.amjhyper.2004.11.002. PMID 15752931
- [Background] Ferrario CM, Basile J, Bestermann W, Frohlich E, Houston M, Lackland DT, Smith RD, Wise DL. The role of noninvasive hemodynamic monitoring in the evaluation and treatment of hypertension. Ther Adv Cardiovasc Dis. 2007 Dec;1(2):113-8. doi: 10.1177/1753944707086095. PMID 19124400
- [Background] Taler SJ. Individualizing antihypertensive combination therapies: clinical and hemodynamic considerations. Curr Hypertens Rep. 2014 Jul;16(7):451. doi: 10.1007/s11906-014-0451-y. PMID 24806735
- [Background] Bour J, Kellett J. Impedance cardiography: a rapid and cost-effective screening tool for cardiac disease. Eur J Intern Med. 2008 Oct;19(6):399-405. doi: 10.1016/j.ejim.2007.07.007. Epub 2008 Feb 11. PMID 18848172
- [Background] Patterson RP. Fundamentals of impedance cardiography. IEEE Eng Med Biol Mag. 1989;8(1):35-8. doi: 10.1109/51.32403. PMID 18238303
- [Background] Cybulski G, Strasz A, Niewiadomski W, Gasiorowska A. Impedance cardiography: recent advancements. Cardiol J. 2012;19(5):550-6. doi: 10.5603/cj.2012.0104. PMID 23042327
- [Background] Cybulski G. Ambulatory impedance cardiography: new possibilities. J Appl Physiol (1985). 2000 Apr;88(4):1509-10. doi: 10.1152/jappl.2000.88.4.1509. No abstract available. PMID 10819621
- [Background] Harvey S, Harrison DA, Singer M, Ashcroft J, Jones CM, Elbourne D, Brampton W, Williams D, Young D, Rowan K; PAC-Man study collaboration. Assessment of the clinical effectiveness of pulmonary artery catheters in management of patients in intensive care (PAC-Man): a randomised controlled trial. Lancet. 2005 Aug 6-12;366(9484):472-7. doi: 10.1016/S0140-6736(05)67061-4. PMID 16084255
- [Background] Richard C, Warszawski J, Anguel N, Deye N, Combes A, Barnoud D, Boulain T, Lefort Y, Fartoukh M, Baud F, Boyer A, Brochard L, Teboul JL; French Pulmonary Artery Catheter Study Group. Early use of the pulmonary artery catheter and outcomes in patients with shock and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2003 Nov 26;290(20):2713-20. doi: 10.1001/jama.290.20.2713. PMID 14645314
- [Background] Tang WH, Tong W. Measuring impedance in congestive heart failure: current options and clinical applications. Am Heart J. 2009 Mar;157(3):402-11. doi: 10.1016/j.ahj.2008.10.016. Epub 2008 Dec 16. PMID 19249408
- [Background] Mills KT, Bundy JD, Kelly TN, Reed JE, Kearney PM, Reynolds K, Chen J, He J. Global Disparities of Hypertension Prevalence and Control: A Systematic Analysis of Population-Based Studies From 90 Countries. Circulation. 2016 Aug 9;134(6):441-50. doi: 10.1161/CIRCULATIONAHA.115.018912. PMID 27502908
- [Background] Polonia J, Martins L, Pinto F, Nazare J. Prevalence, awareness, treatment and control of hypertension and salt intake in Portugal: changes over a decade. The PHYSA study. J Hypertens. 2014 Jun;32(6):1211-21. doi: 10.1097/HJH.0000000000000162. PMID 24675681
- [Background] Nazario Leao R, Marques da Silva P. Diastolic dysfunction in hypertension. Hipertens Riesgo Vasc. 2017 Jul-Sep;34(3):128-139. doi: 10.1016/j.hipert.2017.01.001. Epub 2017 Mar 6. PMID 28268171
- [Background] Krzesinski P, Gielerak GG, Kowal JJ. A "patient-tailored" treatment of hypertension with use of impedance cardiography: a randomized, prospective and controlled trial. Med Sci Monit. 2013 Apr 5;19:242-50. doi: 10.12659/MSM.883870. PMID 23558598
- [Background] Ganau A, Devereux RB, Roman MJ, de Simone G, Pickering TG, Saba PS, Vargiu P, Simongini I, Laragh JH. Patterns of left ventricular hypertrophy and geometric remodeling in essential hypertension. J Am Coll Cardiol. 1992 Jun;19(7):1550-8. doi: 10.1016/0735-1097(92)90617-v. PMID 1534335
- [Background] Nagueh SF, Appleton CP, Gillebert TC, Marino PN, Oh JK, Smiseth OA, Waggoner AD, Flachskampf FA, Pellikka PA, Evangelisa A. Recommendations for the evaluation of left ventricular diastolic function by echocardiography. Eur J Echocardiogr. 2009 Mar;10(2):165-93. doi: 10.1093/ejechocard/jep007. No abstract available. PMID 19270053
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2015 Mar;16(3):233-70. doi: 10.1093/ehjci/jev014. PMID 25712077
- [Background] DeMarzo AP. Using impedance cardiography with postural change to stratify patients with hypertension. Ther Adv Cardiovasc Dis. 2011 Jun;5(3):139-48. doi: 10.1177/1753944711406770. Epub 2011 Apr 28. PMID 21527444
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Derived] Nazario Leao R, Marques Silva P, Branco L, Fonseca H, Bento B, Alves M, Virella D, Palma Reis R. Systolic time ratio measured by impedance cardiography accurately screens left ventricular diastolic dysfunction in patients with arterial hypertension. Clin Hypertens. 2017 Dec 27;23:28. doi: 10.1186/s40885-017-0084-y. eCollection 2017. PMID 29299336